CLINICAL TRIAL: NCT05266807
Title: Fecal Microbiota Transplantation Versus Vancomycin or Fidaxomicin in Clostridioides Difficile Infection First Episode or First Recurrence: A Randomized Controlled, Open-label, Multicenter Phase III Clinical Trial
Brief Title: Fecal Microbiota Transplantation in Clostridioides Difficile Infection First Episode and First Recurrence
Acronym: FENDER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Benoit Guery (Other)
Responsible Party: Sponsor-Investigator, Benoit Guery, Head physician, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FENDER
Record Dates: First submitted 2022-02-18; First posted 2022-03-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides difficile; Clostridium difficile; Fecal Microbiota Transplantation; Vancomycin; Fidaxomicin
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin; Fidaxomicin

STUDY DESIGN:
Intervention Model Description: Randomized, Controlled, Open-label, Multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SoC + oral Fecal Microbiota Transplantation (Experimental): Antibiotic (vancomycin 125 mg 4 times daily or fidaxomicin 200 mg 2 times daily, as initially prescribed per SoC) for 10 days, followed 12h to 4 days later by one oral FMT (20 capsules administered at D1 and 20 capsules at D2), and a second oral FMT if CDI is severe.
  Interventions: Drug: oral capsulized Fecal Microbiota Transplantation; Drug: Vancomycin or Fidaxomicin
- SoC (Active Comparator): Antibiotic (vancomycin 125 mg 4 times daily or fidaxomicin 200 mg 2 times daily, as initially prescribed per SoC) for 10 days.
  Interventions: Drug: Vancomycin or Fidaxomicin

INTERVENTIONS:
Drug: oral capsulized Fecal Microbiota Transplantation — FMT will be administered per os in the form of capsules containing faeces from a healthy donor. Capsules are manufactured at the CHUV pharmacy (University Hospital of Lausanne, Switzerland)
  Arms: SoC + oral Fecal Microbiota Transplantation
Drug: Vancomycin or Fidaxomicin — Vancomycin or Fidaxomicin per os as initially prescribed per SoC

SUMMARY:
The clinical trial aims to evaluate the efficacy of fecal microbiota transplantation (FMT) after standard of care treatment (either vancomycin or fidaxomicin) vs the pragmatic use of standard of care treatment (either vancomycin or fidaxomicin) in severe and non-severe first episode and first recurrence of Clostridioides difficile infection (CDI).

Experimental arm: antibiotic treatment (vancomycin or fidaxomicin as initially prescribed per SoC continued for 10 days) followed by FMT by oral capsules (one FMT, i.e. 20 FMT capsules given on 2 consecutive days, and followed by a 2nd FMT in severe CDI).

Control Arm: vancomycin or fidaxomicin as initially prescribed per SoC continued for 10 days.

DETAILED DESCRIPTION:
Clostridioides difficile (CDI) is well known as major agent of healthcare-associated diarrhea in adult patients. One of the main challenges is the prevention of recurrence of Clostridioides difficile infection which occurs in 15-25% of the cases within the two months following the initial episode. A patient presenting a first recurrence has a higher risk of subsequent recurrences and may enter a cycle of multiple episodes of recurrence leading to significant morbidity, decrease in quality of life, and long courses of antimicrobial therapy. North-American, as well as the European, guidelines propose vancomycin or fidaxomicin to treat this first recurrence. All these recommendations rely on weak to moderate quality of evidence. For patients with multiple recurrences, fecal microbiota transplantation (FMT) is recommended as an option in guidelines based on several randomized controlled trials and a meta-analysis having shown superior efficacy compared to antibiotics with regard to preventing further recurrences.

FMT has never been evaluated for CDI first episode and first recurrence and could represent an attractive treatment to prevent further recurrences, avoid hospitalization (mean length of 10 days) and reduce overall mortality risk.

The aim of our study is to compare the efficacy of FMT (combined with standard treatment: vancomycin or fidaxomicin) compared to standard treatment (vancomycin or fidaxomicin) in patients with a first CDI episode presenting risk factors for recurrence and in patient with a first CDI recurrence.

This is a multicenter, randomized, open-label, phase III superiority trial comparing fecal microbiota transplantation (FMT) delivered via oral capsules after a conditioning standard antibiotic treatment (either vancomycin or fidaxomicin), to the pragmatic use of standard treatment (either vancomycin or fidaxomicin) in non-severe and severe CDI first episode or first recurrence.

Patients (220) will be randomized 1:1. Patients randomized in the FMT arm (Arm A) will continue the antibiotic treatment (vancomycin or fidaxomicin initially prescribed as SoC) for a total of 10 days.

The antibiotic will be stopped for 12h to 4 days and then all patients will receive a first FMT on 2 consecutive days (20 capsules at D1 and 20 capsules at D2). Patients with severe CDI will receive a second FMT immediately administrated at D3 (20 capsules) and at D4 (20 capsules).

Patients randomized in the standard treatment arm (Arm B) will continue the antibiotic treatment (vancomycin or fidaxomicin initially prescribed as SoC) for a total of 10 days.

Efficacy of FMT (combined with standard treatment) will be assessed by comparing the proportion of participants experiencing clinical cure 8 weeks after study treatment completion, in the FMT intervention arm (arm A) and in the standard of care control arm (arm B). Participants will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years old) at the time of informed consent
2. Informed consent signature
3. Medical record documentation of CDI defined as:

   a. A first CDI episode associated with risks factors for recurrence, defined as: i. No CDI episode within the last 8 weeks ii. Current combination of CDI signs and symptoms, confirmed by medical record documentation of microbiological evidence of C. difficile toxin and C. difficile in stools shown by a CDI PCR positive test with Ct < 25 or a toxin A/B EIA positive test and without reasonable evidence of another cause of diarrhea, iii. Presenting at least one of the following risks factors for CDI recurrence:
   * age >65 years-old,
   * hospitalization within the last 3 months,
   * use of proton pump inhibitors (PPI) within the last 3 months,
   * Charlson comorbidity index (CCI) >2,
   * living in long term facility,
   * healthcare- associated CDI (see definition in section 7),
   * severe CDI episode (see definitions in section 6.1.2),
   * immunocompromised patient (except severely immunocompromised according to definitions in section 7.1),
   * history of prior CDI episode(s) (more than 8 weeks ago). OR b. A first CDI recurrence, defined as: i. Previous episode of treated and cured CDI within the last 8 weeks confirmed by medical record documentation of a clinical picture of CDI combined with a positive microbiological CDI test performed according to CDI diagnosis ESCMID guidelines ii. Current combination of CDI signs and symptoms, confirmed by medical record documentation of microbiological evidence of C. difficile toxin and C. difficile in stools shown by a CDI PCR positive test with Ct < 25 or a toxin A/B EIA positive test , and without reasonable evidence of another cause of diarrhea..
4. No multiple episodes (no more than 2 CDI episodes) within 3 last months.
5. Already taking since less than 10 days or will start a course of antibiotics (vancomycin or fidaxomicin) to control recurrent CDI symptoms at the time of screening.
6. Willing and able to have FMT by capsule

Exclusion Criteria:

1. Severe-complicated CDI if at least one of the following signs or symptoms are:

   * ongoing at time of screening and related to CDI: hypotension, septic shock, elevated serum lactate, ileus,
   * or were present at any time of the CDI episode and related to CDI: toxic megacolon, bowel perforation, or any fulminant course of disease (i.e. rapid deterioration of the patient.
2. Prior FMT within 6 months of randomization,
3. Prior colectomy, colostomy, ileostomy, or gastrectomy
4. Metronidazole already given for the treatment of the current CDI for more than 3 days,
5. Need for continued non-anti-CDI systemic antibiotics (should be stopped at randomization at the latest), except prophylactic doses of trimethoprim/sulfamethoxazole,
6. Anticipated indication for antibiotics treatment (for a non-CDI reason) in the next 8 weeks except prophylactic doses of trimethoprim/sulfamethoxazole
7. Other causes of chronic or acute diarrhea beyond CDI (chronic diarrhea is defined as loose/watery stools, which occur three or more times within 24 hours and last for 4 or more weeks)
8. Inflammatory bowel disease,
9. Patients with swallowing disorders, Zenker's diverticulum, gastroparesis, or prior small bowel obstruction,
10. Known hypersensitivity to vancomycin or fidaxomicin,
11. Pregnant/lactating women,
12. Estimated patient's life expectancy of less than 10 weeks,
13. Inability to follow protocol study procedures,
14. Inability to give informed consent,
15. Any condition or medications that will put the participant at greater risk from FMT according to the investigator,
16. Severely immunocompromised
17. No response to anti-CDI antibiotic treatment after at least 5 days of treatment (i.e. no diminution of the daily number of stools at BSS 6-7 compared to first day of treatment; or worsening of CDI severity parameters)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Sustained clinical cure rate | 8 weeks after study treatment completion
  Absence of CDI recurrence through 8 weeks after study treatment completion

SECONDARY OUTCOMES:
Treatment failure | Before 4 weeks and at 5-8 weeks after study treatment completion
  Early and late CDI recurrence rate
CDI new episodes | between 8 weeks and 12 months after study treatment completion
  CDI new episodes occurence rate
Long-term clinical cure | 6 and 12 months after study treatment completion
  Long-term clinical cure rate
Recurrence-free survival rate | 12 months after study treatment completion
  Time from study intervention until CDI recurrence
Overall survival | 12 months after study treatment completion
  Time from study intervention until death
Health status EQ-5D-5L measure (mobility, self-care, usual activities, pain/discomfort, annxiety/depression) | Baseline, 8 weeks, 6 and 12 months after study treatment completion
  5-digit code (score from 1 to 5 for each digit, 1 representing no problem and 5 worse problem)
Health status EQ-5D-5L measure (patient's perception of overall health) | Baseline, 8 weeks, 6 and 12 months after study treatment completion
  EQ Visual Analogue Scale (VAS) score (0 representing the worst health you can imagine to 100 representing the best health you can imagine)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Guery, Principal Investigator — CHUV
Locations (7):
- Switzerland (7):
  - Universitätsspital, Basel, Basel
  - Inselspital Bern, Bern, Canton of Bern
  - HFR Fribourg - Hôpital cantonal, Fribourg, Canton of Fribourg
  - Kantonsspital St Gallen, HOCH, Sankt Gallen, Canton of St. Gallen
  - CHUV, Lausanne, Canton of Vaud
  - Universitätsspital Zürich, Zurich, Canton of Zurich
  - Institut central des hôpitaux, Sion, Valais

IPD SHARING:
Plan to Share IPD: No